CLINICAL TRIAL: NCT03806192
Title: A Field Test of the Partners in Care Program
Brief Title: Feasibility of Partners in Care Program for Caregivers of Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1003619; NCI-2018-03629 (Registry Identifier: NCI / CTRP); 10048 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2020-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Caregiver
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Site intermediary and referring MD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (psychoeducational counseling sessions via telephone) (Experimental): Participants attend 5 psychoeducational counseling sessions over 30-60 minutes via telephone.
  Interventions: Behavioral: Telephone-Based Intervention; Other: Questionnaire Administration
- Group B (psychoeducational counseling sessions in person) (Experimental): Participants attend 5 psychoeducational counseling sessions over 30-60 minutes via video teleconference.
  Interventions: Other: Behavioral, Psychological or Informational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Telephone-Based Intervention — Attend psychoeducational counseling sessions via telephone
  Arms: Group A (psychoeducational counseling sessions via telephone)
Other: Behavioral, Psychological or Informational Intervention — Attend psychoeducational counseling sessions via video teleconference
  Arms: Group B (psychoeducational counseling sessions in person)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies the feasibility of delivering the Partners in Care Program to caregivers of patients with acute myeloid leukemia. Psychological counseling interventions, such as the Partners in Care Program, may help to improve caregivers' psychosocial functioning, marital adjustment in the context of the cancer, communication, and support skills to the patient.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP A: Participants attend 5 psychoeducational counseling sessions over 30-60 minutes via telephone.

GROUP B: Participants attend 5 psychoeducational counseling sessions over 30-60 minutes via video teleconference.

After completion of study, participants are followed up at 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML within the recent 2 months
* Caregivers and patients need to write, read, and speak English as one of their languages of choice; and currently sharing a residence at least 50% of the time together
* Patient must have no other concurrent cancer diagnosis except for basal or squamous cell
* Caregiver must be able to sustain up to 60 minutes of interaction with patient educator
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants will be excluded if either the patient or the caregiver cannot write, read, and speak English as one of their languages of choice; are not currently sharing a residence at least 50% of the time together
* The patient cannot have another concurrent cancer diagnosis except for basal or squamous cell
* Caregiver cannot sustain up to 60 minutes of interaction with the patient educator
* Caregiver does not have access to a computer with 2-way video capability (i.e. ZOOM) or a cell phone

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment | Up to 1 year
Rate of enrollment | Up to 1 year
Rate of completion of 5-session intervention | Up to 1 year

SECONDARY OUTCOMES:
Change in standardized measures of caregiver and patients' scores in each group on anxiety (State-Trait Anxiety Inventory [STAI]) | Baseline up to 4 months
  Will assess the within-group changes using the one-sample t-test or the signed-rank test, as appropriate.
Change in standardized measures of caregiver and patients' scores in each group on depressed mood (Center for Epidemiologic Studies Depression Scale [CES-D]) | Baseline up to 4 months
  Will assess the within-group changes using the one-sample t-test or the signed-rank test, as appropriate.
Change in standardized measures of caregiver and patients' scores in each group on Spouse Skills Checklist | Baseline up to 4 months
  Will assess the within-group changes using the one-sample t-test or the signed-rank test, as appropriate.
Change in standardized measures of caregiver and patients' scores in each group on Cancer Self-efficacy (CASE) | Baseline up to 4 months
  Will assess the within-group changes using the one-sample t-test or the signed-rank test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Lewis, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No